CLINICAL TRIAL: NCT00015704
Title: An Open-Label, Pilot Study Utilizing CD4 T-Cell Counts Lower Than 350 Cells/mm3 as the Threshold for Restarting Therapy With Potent Antiretroviral Therapy With or Without Interleukin-2 to Determine the Effect of Pulse Therapy on the Characteristics of Treatment Interruptions
Brief Title: Effect of Interleukin-2 on HIV Treatment Interruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5102; 10179 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2001-05-01; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Treatment Interruption; Drug Administration Schedule; CD4 Lymphocyte Count; Anti-HIV Agents; Tetanus Toxoid; Aldesleukin; Diphtheria Toxoid
MeSH Terms: conditions — HIV Infections; Tetanus | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
Interleukin-2 (IL-2) helps the body make infection-fighting white blood cells, including CD4 and CD8 T cells. One HIV treatment strategy is planned treatment interruption (stopping anti-HIV drugs when CD4 count and level of virus in the blood are at certain levels). The purpose of this study is to see if IL-2 used with potent anti-HIV drugs allows for longer HIV treatment interruptions.

DETAILED DESCRIPTION:
One approach in reconstituting an HIV-diminished immune system is the use of potent antiretroviral therapy (ART) in conjunction with IL-2. IL-2 is a cytokine secreted by activated T cells that regulates the proliferation and differentiation of CD4 and CD8 T cells. Although treatment with IL-2 can cause temporary increases in HIV viral load, clinical studies with IL-2 have revealed no long-term adverse effects on viral load. IL-2 therapy may also help purge the host's latent viral reservoir through activation of resting lymphocytes harboring provirus. Another approach to managing HIV infection is strategic treatment interruption. Results from small pilot trials suggest that HIV replication can be highly suppressed over consecutive courses of ART following short treatment interruptions, and CD4 T cell counts can be maintained on these interruptions with some positive effect on HIV-specific immunity. This study will evaluate potent ART, started and interrupted based on CD4 cell counts, with or without IL-2.

Patients will be stratified based on lifetime CD4 T-cell nadir (lowest measurement) into one of three groups. Group 1 will have a nadir of 200 CD4 cells/mm3; Group 2 will have a nadir greater than 200 CD4 cells/mm3; and patients with no documented nadir count available will join Group 3. Within each group, patients will be randomly assigned to one of two study arms. Arm A patients will receive pulses of potent ART with IL-2, while Arm B patients will receive pulses of potent ART alone. Patients in Arm A will receive potent ART with IL-2 given by subcutaneous injection twice daily for 5 days every 8 weeks for at least 17 weeks. Arm B patients will receive potent ART alone for at least 17 weeks. Both groups then go on treatment interruption for approximately 64 weeks, followed by potent ART alone for an additional 24 weeks. Patients will repeat this cycle of potent ART with or without IL-2, treatment interruption, and potent ART alone throughout the study. This study will last approximately 4 years.

Clinical and laboratory assessments will be performed periodically throughout the study. CD4 T cell counts and viral load will determine if a patient can enter the next treatment step. Potent ART is not provided by this study.

A5109s is a limited-center substudy designed to determine whether viral replication impairs lymphocyte proliferation in vivo. Patients at substudy-participating sites will register to the substudy immediately after beginning their first treatment interruption in the main study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* On stable, potent ART regimen for at least 3 months prior to study entry
* Viral load of less than 400 copies/ml for at least 6 months prior to study entry
* Viral load of less than 200 copies/ml at screening
* CD4 count of 500 cells/mm3 or greater at screening
* Agree to use acceptable methods of contraception
* Agree to be followed on this study for at least 4 years
* Primary care provider willing to have the patient in the study and to comply with study guidelines

Exclusion Criteria:

* Active or past significant AIDS-related illness. Patients with a history of minimal (less than 10 lesions) cutaneous Kaposi's sarcoma, pulmonary tuberculosis, or bacterial pneumonia are not excluded.
* Immunomodulators within 1 month of study entry
* Hydroxyurea within 3 months of study entry
* Prior IL-2 treatment
* Drugs to treat heart disease within 30 days of study entry
* Serious heart problems
* Cancer requiring anti-cancer drugs
* Thyroid problems. If the condition has been controlled by drugs for at least 3 months prior to study entry, the patient is not excluded.
* Uncontrolled diabetes
* Breathing or stomach problems that, in the opinion of the investigator, may affect the safety of the patient
* History of autoimmune disease, including inflammatory bowel disease, psoriasis, and optic neuritis
* Organ transplant
* History of neurological disorder or mental illness that, in the opinion of the investigator, may interfere with study requirements
* Alcohol or drug abuse that, in the opinion of the investigator, may interfere with study requirements
* Astemizole, midazolam, or triazolam within 2 weeks of study entry
* Systemic corticosteroids for 4 weeks or more within 3 months of study entry
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Keith Henry, MD, Study Chair — HIV Program, Hennepin County Medical Center, University of Minnesota
Locations (17):
- United States (17):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Cornell CRS, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Conrad A. Interleukin-2--where are we going? J Assoc Nurses AIDS Care. 2003 Nov-Dec;14(6):83-8. doi: 10.1177/1055329003255620. PMID 14682072
- [Background] Davey RT Jr, Murphy RL, Graziano FM, Boswell SL, Pavia AT, Cancio M, Nadler JP, Chaitt DG, Dewar RL, Sahner DK, Duliege AM, Capra WB, Leong WP, Giedlin MA, Lane HC, Kahn JO. Immunologic and virologic effects of subcutaneous interleukin 2 in combination with antiretroviral therapy: A randomized controlled trial. JAMA. 2000 Jul 12;284(2):183-9. doi: 10.1001/jama.284.2.183. PMID 10889591
- [Background] Sullivan AK, Hardy GA, Nelson MR, Gotch F, Gazzard BG, Imami N. Interleukin-2-associated viral breakthroughs induce HIV-1-specific CD4 T cell responses in patients on fully suppressive highly active antiretroviral therapy. AIDS. 2003 Mar 7;17(4):628-9. doi: 10.1097/00002030-200303070-00020. PMID 12598786
- [Background] Verheggen R. Immune restoration in patients with HIV infection: HAART and beyond. J Assoc Nurses AIDS Care. 2003 Nov-Dec;14(6):76-82. doi: 10.1177/1055329003259055. PMID 14682071
- [Background] Xu J, Whitman L, Lori F, Lisziewicz J. Methods of using interleukin 2 to enhance HIV-specific immune responses. AIDS Res Hum Retroviruses. 2002 Mar 1;18(4):289-93. doi: 10.1089/088922202753472865. PMID 11860676
- [Result] Henry K, Katzenstein D, Cherng DW, Valdez H, Powderly W, Vargas MB, Jahed NC, Jacobson JM, Myers LS, Schmitz JL, Winters M, Tebas P; A5102 Study Team of the AIDS Clinical Trials Group. A pilot study evaluating time to CD4 T-cell count <350 cells/mm(3) after treatment interruption following antiretroviral therapy +/- interleukin 2: results of ACTG A5102. J Acquir Immune Defic Syndr. 2006 Jun;42(2):140-8. doi: 10.1097/01.qai.0000225319.59652.1e. PMID 16760795
- [Derived] Tebas P, Henry WK, Matining R, Weng-Cherng D, Schmitz J, Valdez H, Jahed N, Myers L, Powderly WG, Katzenstein D. Metabolic and immune activation effects of treatment interruption in chronic HIV-1 infection: implications for cardiovascular risk. PLoS One. 2008 Apr 23;3(4):e2021. doi: 10.1371/journal.pone.0002021. PMID 18431498